CLINICAL TRIAL: NCT01727882
Title: Automated Telephone Follow-up in the Swedish Prison and Probation Services. A Randomized Controlled Trail.
Brief Title: Automated Telephone Follow-up in the Swedish Prison and Probation Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other); Malmö University (Other)
Responsible Party: Principal Investigator, Claes Andersson, PhD, Region Skane
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 535629; 535629 (Other: The Swedish Prison and Probation Services)
Record Dates: First submitted 2012-11-04; First posted 2012-11-16 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Affect; Alcohol Consumption; Substance Abuse
Keywords: Paroled offenders; Interactive Voice Response; Stress; Mental symptoms; Alcohol consumption; Substance use
MeSH Terms: conditions — Alcohol Drinking; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Daily Assessments & Brief Feedback (Experimental): Daily assessments during 30 days after parole and a feedback intervention based on these daily assessments.
  Interventions: Behavioral: Brief feedback; Behavioral: Daily assessments
- Daily assessments (Active Comparator): Daily assessments during 30 days after parole.
  Interventions: Behavioral: Daily assessments

INTERVENTIONS:
Behavioral: Brief feedback — A brief feedback was given on the results of the daily assessments, including a recommendation to the paroled offender and a email report was sent to the probation officer.
  Arms: Daily Assessments & Brief Feedback
Behavioral: Daily assessments — Daily assessment of stress, mental symptoms, alcohol and substance use during 30 consecutive days after parole.

SUMMARY:
The purpose of this study is to investigate whether automated telephony may be used for daily assessments of paroled offenders, and whether a brief intervention based on these daily assessments may result in a more positive development compared to daily assessments only.

DETAILED DESCRIPTION:
To study whether automated telephony could be used in paroled offenders to perform daily assessment of variables associated with recidivism in crime and to study the effects of a brief intervention based on these assessments during 30 days following probation.

ELIGIBILITY:
Inclusion Criteria:

* Convicted criminals subject to parole
* Access to a mobile telephone
* Assigned parole officer at parole

Exclusion Criteria:

* No knowledge of spoken Swedish
* Additional intervention such as intensive supervision with electronic monitoring, or in-patient care at a health and rehabilitation clinic

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2009-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Mental symptoms, SCL-8D | During 30 days after probation
  Mental Symptoms, assessed with SCL-8D (Fink et al. A Nordic multicentre investigation. Part I: Method and prevalence of psychiatric morbidity. Acta Psychiatrica Scandinavica. 1995;92(6):409-418).

SECONDARY OUTCOMES:
Stress | During 30 days after probation
  Stress assessed with the Arnetz and hasson stress questionnaire(Andersson C et al. Measurement properties of the Arnetz and Hasson stress questionnaire in Swedish university freshmen. Scandinavian Journal of Public Health. 2009;37(3):273-279)
Stress | During 30 days after probation
  Daily Assessment of Daily Experience (Stone AA, Neale JM. Development of a methodology for assessing daily experiences. In: Baum A, Singer J, eds. Advances in Environmental Psychology: Environment and Health. Vol 4. New York: Erlbaum; 1982:49-83).
Desire to use alcohol and drugs | During 30 days after probation
  Desire to use alcohol and drugs (Bohn MJ, Krahn DD, Staehler BA. Development and initial validation of a measure of drinking urges in abstinent alcoholics. Alcoholism: Clinical and Experimental Research. 1995;19(3):600-606).
Current use of alcohol and drugs | During 30 days after probation
  Current use was then assessed by simply asking whether the offender had drunk alcohol or used any drugs the previous day.

CONTACTS AND LOCATIONS:
Overall Officials: Claes Andersson, PhD, Principal Investigator — Lund university and Malmö university
Locations (1):
- The Swedish Prison and Probation Services, Region South and Region East, Norrköping, Sweden